CLINICAL TRIAL: NCT01566786
Title: Randomised, Double-Blind, Placebo-Controlled, Multicentre, Dose-Escalation Study to Evaluate the Safety and Preliminary Efficacy of Activated Recombinant Factor VII (NovoSeven®) in Acute Intracerebral Haemorrhage
Brief Title: Safety and Preliminary Efficacy of Activated Recombinant Human Factor VII in Acute Intracerebral Haemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7ICH-1389
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Intracerebral Haemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- activated recombinant human factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — Starting dose of trial drug 10 mcg/kg, escalating up to five dose tiers: 20 mcg/kg, 40 mcg/kg, 80 mcg/kg, 120 mcg/kg and 160 mcg/kg. Administered within the first 4 hours after the insult
  Arms: activated recombinant human factor VII
Drug: placebo — Starting dose of trial drug 10 mcg/kg, escalating up to five dose tiers: 20 mcg/kg, 40 mcg/kg, 80 mcg/kg, 120 mcg/kg and 160 mcg/kg. Administered within the first 4 hours after the insult
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia, Europe and Oceania. The aim of this trial is to evaluate the safety and preliminary efficacy of activated recombinant human factor VII (NovoSeven®) in preventing early haematoma growth in acute Intracerebral Haemorrhage (ICH).

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous ICH diagnosed by CT (Computerized Tomography) scanning within 3 hours of onset
* Signed informed consent form, or in countries where waiver of informed consent is allowed by IRB/IEC, a completed waiver form

Exclusion Criteria:

* Time of onset of symptoms of ICH unknown or more than 3 hours prior to CT
* Patients with secondary ICH related to infarction, haemophilia or other coagulopathy, tumour, trauma, haemorrhagic infarction, cerebrovenous thrombosis, aneurysm, arteriovenous malformations (AVM) or severe trauma
* Surgical haematoma evacuation planned or performed within 24 hours of onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-08; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Change in ICH volume as measured by CT head scans

SECONDARY OUTCOMES:
Occurrence of adverse events
Occurrence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Parkville, Victoria, Australia
- Novo Nordisk Investigational Site, Copenhagen, Denmark
- Novo Nordisk Investigational Site, Jyväskylä, Finland
- Novo Nordisk Investigational Site, Heidelberg, Germany
- Novo Nordisk Investigational Site, Roma, Italy
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Girona, Spain
- Novo Nordisk Investigational Site, Dawan, Taiwan
- Novo Nordisk Investigational Site, Newcastle, United Kingdom

REFERENCES:
- [Result] Mayer SA, Brun NC, Broderick J, Davis S, Diringer MN, Skolnick BE, Steiner T; Europe/AustralAsia NovoSeven ICH Trial Investigators. Safety and feasibility of recombinant factor VIIa for acute intracerebral hemorrhage. Stroke. 2005 Jan;36(1):74-9. doi: 10.1161/01.STR.0000149628.80251.b8. Epub 2004 Nov 29. PMID 15569871
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com